CLINICAL TRIAL: NCT05635344
Title: A Feasibility Window Study of Pembrolizumab Prior to Second Evacuation for Post-molar Gestational Trophoblastic Neoplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C/43/2022; 2022-002986-14 (EudraCT Number)
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Gestational Trophoblastic Disease; Gestational Trophoblastic Neoplasia; Gestational Trophoblastic Tumor, Recurrent
MeSH Terms: conditions — Gestational Trophoblastic Disease; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second evacuation only (No Intervention): Patients that are randomised onto this arm of the study will be treated by second evacuation ALONE.
- Pembrolizumab and second evacuation (Experimental): Patients that are randomised onto this arm will be given a single dose of Pembrolizumab in a neoadjuvant setting followed by second evacuation
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Single dose 200mg dose of Pembrolizumab given intravenously
  Arms: Pembrolizumab and second evacuation

SUMMARY:
Gestational Trophoblastic Diseases (GTD) are a variety of rare, pregnancy related cell multiplication disorders of cells of the placenta which can range from pre-cancerous growths to more serious lesions that can spread to nearby tissues that can cause serious health issues.

Most patients that develop GTD are diagnosed at the precancerous stage early in pregnancy and undergo surgical removal of the disease from the uterus. Around 15% of patients are not cured by surgical removal alone and need to undergo further treatment with chemotherapy or further surgery; of which roughly one-third of patients are cured with a second round of surgery alone.

Anti-cancer treatment with chemotherapy carries many short- and long-term side effects that can negatively affect a person's quality of living. Finding less harmful anticancer therapies that can be paired with surgery is therefore of great benefit to patients with recurrent GTD.

An alternative is to pair surgery with another class of anticancer treatments, known as immunotherapies. Immunotherapy aims to encourage the bodies natural defences to fight the cancer cells.

Pembrolizumab, an immunotherapeutic agent which works by preventing cancer cells from hiding from the immune system; has been proven to be an extremely safe form of anticancer therapy and is an attractive alternative to more toxic chemotherapeutic agents.

The RESOLVE study aims to determine how feasible it is to deliver pre-surgical pembrolizumab to patients and determine if this is a desirable alternative; potentially leading to a larger more definitive study.

20 patients will be recruited onto the study and will be evenly split into two arms:

* 10 patients to receive second evacuation alone
* 10 patients to receive single dose of Pembrolizumab followed by surgery All patients that take part in the study will be recruited from Charing Cross Hospital and will be followed up for a year after the date of their surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to initiation of any study procedures and willingness and ability to comply with the study schedule.
2. Age ≥18yrs
3. Postmolar GTN defined as recurrence or persistence of histologically confirmed CHM after primary surgical evacuation with no intervening treatment.
4. Postmolar GTN defined as plateau or rising human chorionic gonadotropin (hCG). Plateaued hCG is defined as four or more equivalent values of hCG over at least 3 weeks. Rising hCG is defined as two consecutive rises in hCG of 10% or greater over at least 2 weeks.
5. hCG under 20,000 IU/L
6. Low risk disease as defined by the Federation of Obstetrics and Gynecology (FIGO) 2000 risk scoring criteria (score of 6 or less)
7. No metastatic disease on chest X-ray.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
9. Disease present within the uterine cavity not within 5mm of the serosal surface.
10. Adequate bone marrow reserve or organ function as defined by any one of the following parameters:

    * Absolute neutrophil count ≥ 1.5 x 10^9 /L;
    * Platelet count ≥ 100 x 10^9 /L;
    * Haemoglobin ≥ 9.0 g/dL (may have been blood transfused)
    * Creatinine clearance ≥ 30 ml/min (Cockcroft-Gault formula)
    * Serum bilirubin ≤ 1.5 x ULN
    * AST/ALT ≤ 2.5 X ULN
11. All patients must agree to a highly effective method of contraception, or to complete abstinence* for 1 year following second evacuation. This is standard practice following second evacuation of GTN because hCG levels rise in pregnancy thus masking a potential cancer recurrence

Exclusion Criteria:

1. Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, patients who have had any evidence of the other cancer present within the last 2 years or patients whose previous cancer treatment contraindicates this protocol therapy.
2. Patients with histologically confirmed choriocarcinoma, placental site trophoblastic tumor (PSTT) or epithelioid trophoblastic tumor (ETT) on the first curettage.
3. Pregnant women.
4. Uncontrolled vaginal bleeding.
5. Administration of live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. History of immunodeficiency or receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
8. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
9. History of Human Immunodeficiency Virus (HIV) infection.
10. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
11. History of active TB (Bacillus Tuberculosis).
12. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. History of allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of conducting a definitive study of neoadjuvant pembrolizumab prior to second evacuation of low risk postmolar gestational trophoblastic neoplasia (GTN) | 1 year
  Outcome will be measured by determining the proportion of eligible patients who consent to randomisation and the proportion of patients randomised to the intervention arm who complete protocol treatments.
  From this, it can be gauged how feasible it would be to open and recruit to a large scale more definitive study on using pembrolizumab in a neoadjuvant setting in GTN.

SECONDARY OUTCOMES:
To assess the rate of surgical cure with and without pembrolizumab. | 1 year
  Proportion of patients who achieve a sustained complete response (no recurrence of disease) following second evacuation and no further anti-cancer therapy. This defined as normalisation of hCG and no rise by 1 year post procedure. Failure of second evacuation resulting in disease control defined by national guidelines is described as a rise or plateau in hCG, hCG over 20,000 IU/L at 4 weeks or heavy vaginal bleeding. The response rates of patients post second evacuation will be compared across both arms.
To assess the safety of a single dose of pembrolizumab prior to second evacuation versus second evacuation alone. | 12 weeks
  Incidence of adverse effects of second evacuation and pembrolizumab within 30 days and 12 weeks respectively, assessed by Common Terminology Criteria for Adverse Events (CTCAE v5.0, 27 Nov 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Ehsan Ghorani, Study Chair — Imperial College London University
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT05635344/Prot_000.pdf